CLINICAL TRIAL: NCT00750048
Title: Impact of Naloxone on the Analgesic Effect of Paracetamol in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0036
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Pain
Keywords: pain,; sensitization,; analgesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Naloxone; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Naloxone and paracetamol — to check if naloxone induce an inhibiting effect on the analgesic effect of paracetamol in healthy volunteer, using evoked potentials

SUMMARY:
The aim of this study is to check if Naloxone induce an inhibiting effect on the analgesic effect of paracetamol in healthy volunteer, using evoked potentials.

DETAILED DESCRIPTION:
Double Blind, cross-over study in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* between 18 and 40 years old
* written consent given

Exclusion Criteria:

* Naloxone or paracetamol hypersensibility
* Excessive consumption of alcohol, tobacco, coffee, tea or toxicomania
* Concomitant medication

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Variation of amplitude of the N2P2 cerebral wave (before and after administration of Naloxone) induced by thermal stimulus applied on the arm. | before and after administration of Naloxone

SECONDARY OUTCOMES:
Follow up of pain's evaluation using analogical visual scale. Follow up of pain's evaluation using analogical visual scale | following the pain's evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Pickering Gisele, Dr, Principal Investigator — CIC-CPC
Locations (1):
- CPC-CIC, Clermont-Ferrand, France